CLINICAL TRIAL: NCT00386373
Title: Use and Tolerability of Imatinib Mesylate (Gleevec®) in Patients With Philadelphia-Positive Chronic Myeloid or Acute Leukemia During the First 100 Days Following Bone Marrow or Stem Cell Transplantation
Brief Title: Use and Tolerability of Imatinib Mesylate (Gleevec) in Leukemia Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2003-0433
Record Dates: First submitted 2006-10-09; First posted 2006-10-11 (Estimated); Last update posted 2012-08-01 (Estimated); Status verified 2012-07

CONDITIONS: Leukemia
Keywords: Chronic Myeloid Leukemia; CML; ALL; AML; Leukemia; Imatinib Mesylate; Gleevec; Philadelphia-Positive; Bone marrow transplant; BMT; Stem cell transplant; SCT
MeSH Terms: conditions — Leukemia; Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Imatinib Mesylate (Experimental)
  Interventions: Drug: Imatinib Mesylate

INTERVENTIONS:
Drug: Imatinib Mesylate — Starting dose of 100 mg daily by mouth for first 100 days following bone marrow transplant (BMT) or stem cell transplant (SCT).
  Other Names: Gleevec; Imatinib; STI571; NSC-716051

SUMMARY:
Primary Objective:

1. To assess the safety and toxicity of imatinib mesylate when given to patients with Ph (+) CML , ALL or AML within the first 100 days following allogeneic bone marrow or stem cell transplantation.

Secondary Objectives:

1. To identify any clinically significant drug interactions with imatinib in the post-transplant setting.
2. To develop specific monitoring parameters for imatinib use when utilized in the early post-BMT setting.
3. To record one-year survival data in this patient cohort to assess any effect of early imatinib administration on this endpoint.

DETAILED DESCRIPTION:
Imatinib mesylate is an FDA-approved, commercially available drug for patients with acute or chronic leukemias carrying the Philadelphia chromosome. Women who are able to have children must have a negative blood pregnancy test before taking this drug

No earlier than three weeks after the bone marrow or stem cell transplant, you will start taking imatinib mesylate by mouth. You will take it once or twice a day until roughly 100 days following the transplant or until you are released from the Houston area by your M. D. Anderson physician. Imatinib mesylate should be taken with a meal and a glass of water, preferably in the morning.

The dose will be gradually increased as long as you don't experience severe side effects. If severe side effects occur, imatinib will be stopped, either temporarily or permanently.

After about 100 days (or after leaving Houston) the medication may be continued at the discretion of the study doctor, but the study will be considered completed.

This is an investigational study. A total of up to 40 patients will take part in this study. All will be enrolled at M. D. Anderson. The study is partially funded by the manufacturer of imatinib mesylate (see below), although the drug is not provided free of charge.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with Ph(+) CML and/or CML with bcr-abl rearrangement and diploid cytogenetics not eligible for protocols of higher priority (e.g. ID02-901, DM99-081, DM97-206, etc).
2. The disease must be beyond first chronic phase according to IBMTR criteria (i.e. accelerated phase, blastic phase, second chronic phase) at the time of transplant.
3. Patients with Ph(+) acute lymphocytic (or myeloid) leukemia.
4. Patients with diploid cytogenetics but molecular evidence of bcr-abl rearrangement are also eligible.
5. Age >/= 16 years
6. Unsupported ANC at least 1500 and unsupported platelet count of at least 50K following BMT.
7. Patients may have received prior chemotherapy for their disease or be previously untreated.
8. Patients must have received an allogeneic bone marrow or stem cell transplant. Allogeneic transplant types may include matched sibling donors, mismatched related donors, or unrelated donors. All preparative regimens acceptable.
9. Signed informed consent
10. Zubrod status </= 3
11. Adequate hepatic (bilirubin </= 3 mg/dl, transaminases < 4 x upper limit of normal) and renal function (serum creatinine </= 3 mg/dl )

Exclusion Criteria:

1. Grade III/IV cardiac problems as defined by the NYHAC
2. History of hypersensitivity to imatinib
3. Pregnant and lactating women
4. HIV positive

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2003-08; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Toxicity Rate | 100 Days and 1 Year

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Anderlini, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- U.T.M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org